CLINICAL TRIAL: NCT03821363
Title: Recombinant Humanized Anti- PD-1 Monoclonal Antibody（SCT-I10A） in Patients With Advanced Solid Tumors or Lymphoma :a Phase Ⅰ, Open-label, Multicenter Study
Brief Title: Safety, Tolerability, Pharmacokinetics and Efficacy of SCT-I10A in Patients With Advanced Solid Tumors or Lymphoma
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sinocelltech Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: SCT-I10A-X101
Record Dates: First submitted 2019-01-24; First posted 2019-01-29 (Actual); Last update posted 2019-01-29 (Actual); Status verified 2018-07

CONDITIONS: Advanced Solid Tumors or Lymphoma
Keywords: Neoplasms; Solid Tumors; Lymphoma; PD-1; SCT-I10A
MeSH Terms: conditions — Lymphoma; Neoplasms

STUDY DESIGN:
Intervention Model Description: Groups of participants are assigned to receive interventions based on prior milestones being reached in the study, such as in some dose escalation and adaptive design studies
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Low dose group (Experimental): SCT-I10A will be administered at a dose of 60mg, Q3W up to 24 months.
  Interventions: Biological: SCT-I10A
- Middle dose group (Experimental): SCT-I10A will be administered at a dose of 200mg, Q3W up to 24 months.
  Interventions: Biological: SCT-I10A
- High dose group (Experimental): SCT-I10A will be administered at a dose of 600mg, Q3W up to 24 months.
  Interventions: Biological: SCT-I10A

INTERVENTIONS:
Biological: SCT-I10A — Experimental: Anti- PD-1 monoclonal antibody（SCT-I10A）

SUMMARY:
The purpose of this study is to evaluate the safety, tolerability, pharmacokinetics and preliminary efficacy of recombinant humanized anti- PD-1 monoclonal antibody（SCT-I10A）in patients with advanced solid tumors or lymphoma treated after failure of standard therapy.

DETAILED DESCRIPTION:
This open label, multicenter phase I study is designed to evaluate the safety, tolerability, pharmacokinetics and preliminary efficacy in advanced solid tumors or lymphoma treated with anti- PD-1 monoclonal antibody SCT-I10A. The trial will be divided into two parts: dose-exploration and indication expansion.

ELIGIBILITY:
Inclusion Criteria:

* Able to provide written informed consent before screening；
* Males or females. Aged 18 to 75 years old;
* Life expectancy≥12 weeks before starting treatment (clinical assessment);
* With an Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1;
* Histologically or cytologically confirmed advanced solid tumor or lymphoma;
* Advanced solid tumor or lymphoma with standard treatment failed or no effective therapy;
* According to RECIST 1.1 or Lugano 2014 criteria, patients must have at least one measurable lesion that can be accurately assessed;
* Adequate organ and bone marrow function as defined below:

Absolute neutrophil count (ANC) greater than/equal to 1.5×l09/L; Platelets greater than/equal to 75×109/L; Hemoglobin greater than/equal to 80g/L; Aspartate aminotransferase (AST)/alanine aminotransferase (ALT) less than/equal to 2.5 times ULN, or less than/equal to 5 times ULN if known liver metastases; Total bilirubin less than/equal to 1.5 times ULN; Serum creatinine less than/equal to 1.5 times ULN or Ccr>50ml/min; Thyroid stimulating hormone (TSH) hormone levels less than/equal to ULN.

Exclusion Criteria:

* Patients who are allergic to analogue of SCT-I10A and/or its inactive ingredients;
* Patients have been treated with anti-PD-L1 and anti-PD-1 antibody;
* Patients are currently enrolled in other research devices or in research drugs, or less than 4 weeks from other research drugs or devices;
* Within 4 weeks prior to the first dose of study drug, patients have received anti-tumor drugs (such as chemotherapy, endocrine therapy, targeted therapy, immune therapy, tumor embolization). Within 6 weeks prior to the first dose of study drug, patients have been treated with biological products, nitrosourea or mitomycin C;
* Within 2 weeks prior to the first dose of study drug, patients have received corticosteroids or other immunosuppressive agents;
* Within 4 weeks prior to the first dose of study drug, patients have received live attenuated vaccine (LAV), or who planned to use LAV during the study period;
* Within 4 weeks prior to the first dose of study drug, patients have received major surgery, or had wounds, ulcers or fractures that haven't healed;
* Prior to the first dose of study drug, patients had toxicity due to previous anti-tumor treatment, which hasn't return to Grade 0-1 according to the NCI CTCAEv4.03;
* Patient with cerebrospinal meningitis metastasis or central nervous system metastasis with untreated or uncontrolled with other treatment;
* Patients with an active, known or suspected autoimmune disease or a history of autoimmune disease;
* Patients with a history of allogeneic organ transplantation or allogeneic hematopoietic stem cell transplantation;
* Within 6 months prior to study, patients had uncontrolled concurrent diseases, including but not limited to acute myocardial infarction, unstable angina pectoris, stroke, or transient ischemic attack, congestive heart failure (NYHA, greater than II), left ventricular ejection fraction (LVEF) <50%, and with related heart disease. Patients with chronic or acute disease, psychological or psychiatric disorders, laboratory abnormalities which may affect subject compliance and outcomes in this clinical study;
* Patients with HIV, active hepatitis B (HBV DNA≥104 copies/ml) or active hepatitis C (HCV RNA≥103 copies/ml), etc.;
* Patients who have interstitial lung disease, such as interstitial pneumonia, pulmonary fibrosis, or CT or MRI reminder ILD.
* Patients with clinical symptoms, required clinical intervention or stable time less than 4 weeks of serous cavity effusion (such as pleural effusion and ascites);
* Patients with other primary malignancies;
* Pregnant or lactating women;
* Patients who were not willing to accept effective contraceptive measures during treatment and within 6 months after treatment;
* Subjects who are considered not suitable for the study by investigator.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 206 (Estimated)
Dates: Start 2018-12-13 (Actual); Primary Completion 2020-07 (Estimated); Study Completion 2020-07 (Estimated)

PRIMARY OUTCOMES:
Safety/Tolerability | 24 months
  Incidence of adverse events and outlier of laboratory tests, positive rate of immunogenicity

SECONDARY OUTCOMES:
Objective response rate (ORR) | 24 months
  ORR is defined as proportion of patients achieving complete response (CR) or partial response (PR) according to RECIST v1.1 or Lugano 2014 criteria during trial treatment.
Duration of response (DOR) | 24 months
  DOR is defined as time from the date when a patient first meets the criteria for CR or PR according to RECIST v1.1 or Lugano 2014 criteria, until the date that progressive disease (PD) is objectively documented or death, whichever occurs first.
Disease control rate (DCR) | 24 months
  PFS is defined as the time from first dose of SCT200 until the date of first documentation of progression or date of death, whichever occurs first,according to RECIST v1.1 or Lugano 2014 criteria.
Progression free survival (PFS) | 24 months
  PFS is defined as the time from first dose of SCT200 until the date of first documentation of progression or date of death, whichever occurs first,according to RECIST v1.1 or Lugano 2014 criteria.
Overall survival (OS) | 24 months
  OS is defined as time from first dose of SCT200 until the date of death from any cause.

CONTACTS AND LOCATIONS:
Locations (1):
- The Fifth Medical Center of PLA General Hospital, Beijing, Beijing Municipality, China